CLINICAL TRIAL: NCT03258801
Title: Pirfenidone as Bridging Therapy for Lung Transplant in Patients Suffering From Idiopathic Pulmonary Fibrosis
Status: Withdrawn | Type: Observational
Why Stopped: Clinical evaluation plan outdated and obsolete due to altered clinical routine
Sponsor: Dr. Christopher Lambers (Other)
Collaborators: Clinical Trials Coordination Centre, Medical University of Vienna (Unknown)
Responsible Party: Sponsor-Investigator, Dr. Christopher Lambers, Ass. Prof., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: NIS-ML-29952
Record Dates: First submitted 2017-08-18; First posted 2017-08-23 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Idiopathic Pulmonary Fibrosis; Lung Transplant; Complications
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pirfenidone: Patients who are admitted to the lung transplantation department and fulfill the international criteria for idiopathic pulmonary fibrosis and are treated with Pirfenidone as bridging therapy.
- Control: Patients who are admitted to the lung transplantation department and fulfill the international criteria for idiopathic pulmonary fibrosis and are not treated with Pirfenidone.

SUMMARY:
The diagnosis of idiopathic pulmonary fibrosis (IPF) is currently one of the most common diagnoses for patients under evaluation for lung transplantation. In recent years, an absolute increase in prevalence/ incidence of IPF has been observed. There is evidence that patients with IPF on waiting list for lung transplantation might benefit from pirfenidone treatment. Until now, no data are published regarding this important issue in lung transplantation.

Primary objective is to determine whether there is a difference in the duration time of mechanical ventilation (weaning) directly after lung transplantation between patients treated with pirfenidone and patients without pirfenidone treatment. The Secondary objectives are to determine whether there are differences between the pirfenidone treatment group and the control group regarding survival after LUTX, the score on the Saint Georges Respiratory Questionnaire and the decline in forced vital capacity (FVC%) In this Investigator initiated, non- interventional single center study , patients on the waiting list for transplant pirfenidone treatment receive oral pirfenidone at the standard dose of 2403 mg per day. The treatment duration will range from 6 to 12 months. A control group will be used to correlate the outcome-parameters for a descriptive comparison. The control group includes patients with IPF on the waiting list who were on another IPF specific (or no) treatment for IPF The Study Population are Patients aged between 40-70 years who are admitted to the lung transplantation department and fulfill the international criteria for idiopathic pulmonary fibrosis ( existence of a usual interstitial pneumonia (UIP) pattern in the high-resolution computed tomography (HRCT) is necessary).

Variables: Duration of mechanical ventilation after LUTX (hours), Forced Vital capacity relative to reference value at baseline (FVC0%), Forced Vital capacity relative to reference value after 6 months (FVC6%),Forced Vital capacity relative to reference value after 12 months (FVC12%) Study Size: 30 patients in the Pirfenidone group, 20 patients in the control group.

For the primary Endpoint, the mean, standard deviation, median, minimum and maximum of the weaning time of patients who received a pirfenidone treatment, as well as of patients from the control group will be computed and presented in a table. Additionally, a Kaplan-Meier curve will be estimated and plotted alongside the respective 95% CI calculated using the method of Brookmeyer and Crowley. Furthermore, a stepwise linear regression using forward selection and Age, RBMI, FVC0%, (FVC6%-FVC0%), TLC, FEV1% and ECMO, as well as the pirfenidone treatment as predictors will be computed. The null hypothesis is that the pirfenidone treatment has no influence on the weaning time. The according model coefficient estimate and standard error will be used to test the null hypothesis using a t-test at significance level α=0.05.

For the secondary endpoints, the mean, standard deviation, median, minimum and maximum of patients who received a pirfenidone treatment, as well as of patients from the control group will be computed and presented in a tableStepwise Cox Regression using forward selection and Age, RBMI, FVC0%, (FVC6%-FVC0%) and ECMO, as well as the pirfenidone treatment as predictors will be computed in order to compare the treatment and the control group a . If p-values are calculated for the secondary endpoint analysis, they serve only descriptive purposes. Therefore no multiple testing corrections are applied.

ELIGIBILITY:
Inclusion Criteria:

For Pirfenidone Group

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study

* mild to moderate idiopathic pulmonary fibrosis (IPF).
* Current or intended treatment with Pirfenidone
* Diagnosis of Interstitial Lung disease
* Evaluation for Lung Transplantation
* Age 40-70

For Control Group

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study

* mild to moderate idiopathic pulmonary fibrosis (IPF).
* Diagnosis of Interstitial Lung disease
* Evaluation for Lung Transplantation
* Age 40-70

Exclusion Criteria:

For Pirfenidone Group

* Other lung diseases (such as cystic fibrosis, COPD)
* Infection with Hepatitis C,
* Liver cirrhosis CHILD C
* Coronary heart disease (3VD)

For Control Group

* Other lung diseases (such as cystic fibrosis, COPD)
* Infection with Hepatitis C,
* Liver cirrhosis CHILD C
* Coronary heart disease (3VD)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are admitted to the lung transplantation department and fulfill the international criteria for idiopathic pulmonary fibrosis will be evaluated (existence of a usual interstitial pneumonia (UIP) pattern in the high-resolution computed tomography (HRCT) is necessary).
  The assignment of a patient to a particular therapeutic strategy remains in the sole responsibility of the treating physician and must not be dictated by this study-specific observation- and evaluation plan
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Duration time of mechanical ventilation (weaning) directly after lung transplantation | First two weeks after lung transplantation
  Duration of mechanical ventilation after LUTX measured in days

SECONDARY OUTCOMES:
Days of survival after LUTX | First 90 days after LUTX
  Days of survival after LUTX measured in days
decline in forced vital capacity (FVC%) from baseline to 6 months | from baseline to 6 months
  decline in forced vital capacity (FVC%) from baseline to 6 months
decline in forced vital capacity (FVC%) from baseline to 12 months | from baseline to 12 months
  decline in forced vital capacity (FVC%) from baseline to 12 months
decline in forced vital capacity (FVC%) from 6 months to 12 months | from 6 months to 12 months
  decline in forced vital capacity (FVC%) from 6 months to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Department of Surgery, Vienna, Austria